CLINICAL TRIAL: NCT02472873
Title: Efficacy of Aspiration and Sclerotherapy During Laparoscopy Using 95% Ethanol for the Treatment of Endometriomas - a Prospective Case Control Study
Brief Title: Efficacy of Aspiration and Sclerotherapy During Laparoscopy Using 95% Ethanol for the Treatment of Endometriomas
Acronym: EASLETE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Dana Josephy, Dr., Meir Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0062-15
Record Dates: First submitted 2015-06-07; First posted 2015-06-16 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Endometrioma; Endometriosis
Keywords: endometrioma; endometriosis; sclerotherapy; ethanol; aspiration; laparoscopy
MeSH Terms: conditions — Endometriosis | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- study group - sclerotherapy (Experimental): Aspiration and Sclerotherapy of endometriomas.
  Interventions: Procedure: Aspiration and Sclerotherapy of endometriomas.; Drug: Ethanol
- control group - cystectomy (Other): cystectomy of endometriomas.
  Interventions: Procedure: cystectomy of endometriomas.

INTERVENTIONS:
Procedure: Aspiration and Sclerotherapy of endometriomas. — Aspiration and Sclerotherapy During Laparoscopy Using 95% Ethanol for the Treatment of Endometriomas
  Arms: study group - sclerotherapy
Procedure: cystectomy of endometriomas. — cystectomy of endometriomas during laparoscopy
  Arms: control group - cystectomy
Drug: Ethanol
  Arms: study group - sclerotherapy

SUMMARY:
The purpose of this study is to evaluate the efficacy of aspiration and sclerotherapy during laparoscopy using 95% ethanol for the treatment of endometriomas, compared to the standard cystectomy treatment - a prospective case control study.

DETAILED DESCRIPTION:
Women who are candidates for elective laparoscopy for the treatment of ovarian ensometriomas will be assigned to one of two groups - a) standard cystectomy treatment, b) aspiration and sclerotherapy using 95% ethanol. The women will be introduced with both operative options and they will choose which one they prefer. After an elaborate explanation about the study they will sign an informed consent form. the following data will be collected prior the operation: age, gravity & parity, operative history, general medical history, the cyst size, AMH (Anti Mullerian Hormone), AFC (Antral Follicle Count), symptoms related to endometriosis (through a questionnaire), fertility history including any fertility treatment in the past and planned pregnancy after the operation.

The laparoscopy will take place in Meir Medical Center. in the study group the cyst content will be aspirated and flushed with normal saline. 95% sterile ethanol will be instilled into the cyst through a foley catheter. Ethanol will be left in the cyst for a maximum of 15 min then aspirated as completely as possible following normal saline flushing. In the control group we will follow the standard treatment which is cystectomy.

The women will be followed 4 and 6 months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* women with endometrial cyst ≥ 4 cm.
* candidates for elective laparoscopy due to endometriosis.
* age 18-45 years

Exclusion Criteria:

* endometrial cyst < 4 cm.
* an emergency surgery.
* age <18 or >45
* women with a history of tubal ovarian abscess (TOA).
* high index of suspision for ovarian malignancy.
* ethanol sensitivity.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-06; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
endometrioma recurrence rate | up to 6 months after the laparoscopy
  Ultrasound examination that demonstrate the presence/lack of ovarian cyst with sonographic features of endometrioma in the ovary where the sclerotherapy took place.

SECONDARY OUTCOMES:
length of surgery | intraoperative
  the time from insertion of the first trocar until closing of the abdominal wall.
length of hospital stay | participants will be followed for the duration of hospital stay, an expected average of 2 days
complication rate | during the surgery and until one month after the surgery.
  infection, excessive bleeding, injury to other abdominal organs
Measure of efficacy of the treatment by questionnaire | 4 months and 6 months after the laparoscopy
Ovarian reserve | 4 months and 6 months after the laparoscopy
  Anti mullerian hormone (AMH) and antral follicle count (AFC) measurement 4 months and 6 months after the laparoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Dana Josephy, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir medical center, Kfar Saba, Israel

REFERENCES:
- [Background] Koike T, Minakami H, Motoyama M, Ogawa S, Fujiwara H, Sato I. Reproductive performance after ultrasound-guided transvaginal ethanol sclerotherapy for ovarian endometriotic cysts. Eur J Obstet Gynecol Reprod Biol. 2002 Oct 10;105(1):39. doi: 10.1016/s0301-2115(02)00144-6. PMID 12270563
- [Background] Suganuma N, Wakahara Y, Ishida D, Asano M, Kitagawa T, Katsumata Y, Moriwaki T, Furuhashi M. Pretreatment for ovarian endometrial cyst before in vitro fertilization. Gynecol Obstet Invest. 2002;54 Suppl 1:36-40; discussion 41-2. doi: 10.1159/000066293. PMID 12441659
- [Background] Chapron C, Vercellini P, Barakat H, Vieira M, Dubuisson JB. Management of ovarian endometriomas. Hum Reprod Update. 2002 Nov-Dec;8(6):591-7. doi: 10.1093/humupd/8.6.591. PMID 12498427
- [Background] Shaw RW. Treatment of endometriosis. Lancet. 1992 Nov 21;340(8830):1267-71. doi: 10.1016/0140-6736(92)92960-n. No abstract available. PMID 1359330
- [Background] Busacca M, Chiaffarino F, Candiani M, Vignali M, Bertulessi C, Oggioni G, Parazzini F. Determinants of long-term clinically detected recurrence rates of deep, ovarian, and pelvic endometriosis. Am J Obstet Gynecol. 2006 Aug;195(2):426-32. doi: 10.1016/j.ajog.2006.01.078. PMID 16890551
- [Background] Zanetta G, Lissoni A, Dalla Valle C, Trio D, Pittelli M, Rangoni G. Ultrasound-guided aspiration of endometriomas: possible applications and limitations. Fertil Steril. 1995 Oct;64(4):709-13. doi: 10.1016/s0015-0282(16)57843-1. PMID 7672139
- [Background] Akamatsu N, Hirai T, Masaoka H, Sekiba K, Fujita T. [Ultrasonically guided puncture of endometrial cysts--aspiration of contents and infusion of ethanol]. Nihon Sanka Fujinka Gakkai Zasshi. 1988 Feb;40(2):187-91. Japanese. PMID 3283269
- [Background] Kafali H, Yurtseven S, Atmaca F, Ozardali I. Management of non-neoplastic ovarian cysts with sclerotherapy. Int J Gynaecol Obstet. 2003 Apr;81(1):41-5. doi: 10.1016/s0020-7292(02)00401-0. PMID 12676392
- [Background] Bret PM, Atri M, Guibaud L, Gillett P, Seymour RJ, Senterman MK. Ovarian cysts in postmenopausal women: preliminary results with transvaginal alcohol sclerosis. Work in progress. Radiology. 1992 Sep;184(3):661-3. doi: 10.1148/radiology.184.3.1509048.
- [Background] Noma J, Yoshida N. Efficacy of ethanol sclerotherapy for ovarian endometriomas. Int J Gynaecol Obstet. 2001 Jan;72(1):35-9. doi: 10.1016/s0020-7292(00)00307-6. PMID 11146075
- [Background] Hsieh CL, Shiau CS, Lo LM, Hsieh TT, Chang MY. Effectiveness of ultrasound-guided aspiration and sclerotherapy with 95% ethanol for treatment of recurrent ovarian endometriomas. Fertil Steril. 2009 Jun;91(6):2709-13. doi: 10.1016/j.fertnstert.2008.03.056. Epub 2008 Jun 20. PMID 18571165
- [Background] Takuma N, Sengoku K, Pan B, Wada K, Yamauchi T, Miyamoto T, Ohsumi D, Ishikawa M. Laparoscopic treatment of endometrioma-associated infertility and pregnancy outcome. Gynecol Obstet Invest. 2002;54 Suppl 1:30-4; discussion 34-5. doi: 10.1159/000066292. PMID 12441658